CLINICAL TRIAL: NCT01493895
Title: Study Assessing Safety and Efficacy of B-cure Laser Treating Diabetic Chronic Wounds
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: becure-CTIL-HMO
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2013-03-22 (Estimated); Status verified 2013-03

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group, (Active Comparator): The control group will be treated with a sham B-cure laser machine, emitting only green indicator light and no 808nm laser.
  Interventions: Device: standard hoem treatment
- study, LLLT-808 B-cure laser machine (Experimental): The study group will be treated with the LLLT-808 B-cure laser machine, emitting the 808nm laser beam together with a green indicator light.
  Interventions: Device: LLLT-808 B-cure laser machine

INTERVENTIONS:
Device: standard hoem treatment — All treatments will be carried out by trained study caregivers that will give standard treatment to all the participants under their care.
  Every treatment will consist of the following steps:
  A thorough rinse with an antiseptic soap (Septal scrub) with a stream of warm water.
  Drying of the foot with an absorbable disposable paper towel. Using clean latex gloves the caregiver will beam the ulcer with LLLT 808, B-cure laser machine in the following method.
  Arms: control group,
Device: LLLT-808 B-cure laser machine — From the day of entering the study, ulcers will be treated twice daily regardless of the treatment that was used until then.
  All treatments will be carried out by trained study caregivers that will give standard treatment to all the participants under their care.
  Every treatment will consist of the following steps:
  A thorough rinse with an antiseptic soap (Septal scrub) with a stream of warm water.
  Drying of the foot with an absorbable disposable paper towel. Using clean latex gloves the caregiver will beam the ulcer with LLLT 808, B-cure laser machine in the following method.
  The part of the laser machine from which the laser beam is radiating - the beam guard, will be cleaned with a disposable swab of 70% alcohol. The cleaning will be performed while the machine is pointing downwards.
  Arms: study, LLLT-808 B-cure laser machine

SUMMARY:
For centuries, light has been a well-known and effective healing method. In the beginning of the 20th century there was a first attempt to condense light energy and distribute it in higher levels, a use that was successfully applied on many soldiers wounded in the Second World War. The laser, which is based on the quantum phenomenon of stimulated emission, was first demonstrated in the beginning of the 1960s and immediately received many applications in all areas of medicine.Many different studies were carried out in the past decade trying to assess the effect of laser therapy on properties of healing wounds. This study aim to assess the efficacy and safety of Low-Level Laser Therapy (LLLT) in the treatment of non-healing diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Known Diabetes mellitus
2. With an active chronic wound in the foot, that has been treated conventionally for over 3 months.
3. No known osteomyelitis.
4. Size of wound: 1-8 cm2.
5. Ages: 21 - 75
6. Gender: male and female

Exclusion Criteria:

1. Signs of osteomyelitis.
2. The ability to probe to bone with the presence of local or systemic infection and suggestive radiological features provided a clinical diagnosis of osteomyelitis.
3. There is active osteomyelitis in the bone underlying the ulcer.
4. Pregnant women.
5. Children under 21.
6. Presence of or known cancerous comorbidity.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To assess the efficacy of b-cure laser in patients with diabetes mellitus induced lower leg skin ulcers
  the efficacy will be assesed using measurement of wound depth.

SECONDARY OUTCOMES:
safety
  safety will be evaluated by counting advese events in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Haze A, Gavish L, Elishoov O, Shorka D, Tsohar T, Gellman YN, Liebergall M. Treatment of diabetic foot ulcers in a frail population with severe co-morbidities using at-home photobiomodulation laser therapy: a double-blind, randomized, sham-controlled pilot clinical study. Lasers Med Sci. 2022 Mar;37(2):919-928. doi: 10.1007/s10103-021-03335-9. Epub 2021 May 29. PMID 34052927